CLINICAL TRIAL: NCT00994435
Title: The Incretin Secretion in the Gut System Related to the Physiological Stimulus
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Ghirlanda G. MD, Catholic University of the Sacred Heart
Other Study IDs: 1082/08
Record Dates: First submitted 2009-10-01; First posted 2009-10-14 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2009-10

CONDITIONS: Obesity
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Insulin secretion and insulin sensitivity are related with an inverse, hyperbolic function, the so called disposition index, that shows the critical importance of the ß-cell dysfunction for the development of T2DM. A consequence of the hyperbolic relationship is that increased insulin resistance is compensated by up-regulation of insulin secretion, as it happens in obesity. However, when a defective insulin secretion in relation to insulin sensitivity takes place (i.e. reduced disposition index) then impaired glucose tolerance or type 2 diabetes develop. The investigators have recently demonstrated that bilio-pancreatic diversion determines a prompt reversibility of T2DM by normalizing peripheral insulin sensitivity and enhancing ß-cell sensitivity to glucose; these changes occur within few days after surgery, largely before changes in body weight occur. This operation may affect the entero-insular axis function, by diverting nutrients away from the proximal gastro-intestinal tract and by delivering incompletely digested nutrients to the ileum, thus abnormally stimulating the secretion of intestinal incretins. It has been shown that male Wistar rats undergoing three different types of small intestinal surgery, namely ileal transposition (either 10 or 20 cm of lower ileum transposed to mid-duodenum) or 85% jejuno-ileal bypass, showed a sustained post-operative reduction in food intake and a significant change in body weight gain. All experimental groups had a large increase in basal and meal-stimulated enteroglucagon, while the area under the curve of plasma levels of gastrin, gastric inhibitory polypeptide (GIP), insulin and blood glucose were significantly reduced. GIP is produced mainly in the duodenum and jejunum as shown in dogs .The aim of the present study is to investigate the intestinal site of production of incretins in response to intraluminal nutrients stimulation in order to establish the relationship between insulin resistance, insulin hypersecretion and different small intestinal segments in insulin resistance conditions, such as obesity and T2DM. To this purpose a mixed test meal will be infused in the duodenum, proximal jejunum or ileum and glucose uptake and insulin secretion studied, in relation to glucagon and incretin response. Studies are carried out in 20 obese subjects of both sexes, 10 of whom with type 2 diabetes and 10 with normal glucose tolerance.

DETAILED DESCRIPTION:
For intestinal perfusion, a tube assembly (outer diameter 7 mm) marked with a length scale is used. It consists of six tubes that are bonded together with tetrahydrofuran (Sigma Chemical Corp, St Louis, Missouri, USA). Three tubes are connected to a balloon which is used to occlude the intestinal lumen proximal to the site of infusion. Three tubes are radio-opaque to allow fluoroscopic location of the assembly; their distal end is immediately distal to the proximal occluding balloon(perfusion site) and positioned at 60 cm (duodenum), 90 cm (proximal jejunum) and 120 cm (distal jejunum) from the nose. After a 12 hour fast, the subjects swallow the tube assembly. The position of the assembly is confirmed by fluoroscopy. With the tube in the right position, the occluding balloon is inflated with 60 ml of air and perfusion of the distal intestinal segment is started. . The perfusion is performed using a continuous pump according to the following scheme:

100 ml/h during 30 minutes 110 ml/h during 60 minutes 123 ml/h during 60 minutes 133 ml/h during 30 minutes test period, which is followed by 120 minute absorption period. Each subject will be studied in 3 different sessions at 7-10 days distance randomly selected in order to study the effect on insulin sensitivity and secretion of a test meal delivery in different intestinal segments (i.e. at the duodenum, the proximal jejunum, and the distal jejunum). Blood samples for glucose, free fatty acids (FFA) insulin, C-peptide, glucagon, GLP-1, GIP, are drawn at -30 minutes and at 0, 15, 30, 40, 60, 80, 100, 120, 150, 180, 240, 300 and 360 minutes during each of the test periods. The lipid-glucose-protein test meal is a mixture of ScandiShake(85 g of powder is mixed in 240-mL milk resulting in 69.5 g carbohydrates, 30.4 g fat, and 11.7 g protein).

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Women in fertile age should engage themselves in avoiding pregnancy during the study protocol. Before starting each experimental session a pregnancy test will be performed and pregnant women excluded from the investigation. All women will be studied in the follicular phase of their menstrual cycle 30 to 60 years old.
* HbA1c between 6.5 and 8.5% (for patients with T2DM only)
* BMI between 30-40 Kg /m2

Exclusion Criteria:

* Past or active medical history of major endocrinological, renal, cardiac, respiratory, liver or gastro-intestinal diseases.
* All Diabetic patients must have never been treated with oral hypoglycemic agents or insulin.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Studies are carried out in 20 obese subjects of both gender sexes, 10 of whom with type 2 diabetics and 10 with normal glucose tolerance.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
dosage for glucose, free fatty acids (FFA) insulin, C-peptide, glucagon, GLP-1, GIP | 3 test meals of 360 minutes duration each, taken at a time distance of 7-10 days . Overall duration, approximally 30 days for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ghirlanda, MD, Principal Investigator — Catholic University
Locations (1):
- Department of Metabolic Diseases, Institute of Internal Medicine - Catholic University, Rome, Rome, Italy

REFERENCES:
- [Derived] Salinari S, Carr RD, Guidone C, Bertuzzi A, Cercone S, Riccioni ME, Manto A, Ghirlanda G, Mingrone G. Nutrient infusion bypassing duodenum-jejunum improves insulin sensitivity in glucose-tolerant and diabetic obese subjects. Am J Physiol Endocrinol Metab. 2013 Jul 1;305(1):E59-66. doi: 10.1152/ajpendo.00559.2012. Epub 2013 May 7. PMID 23651846